CLINICAL TRIAL: NCT04428437
Title: An Observational Study to Evaluate the Safety and Efficacy of Lenvatinib in HCC Subjects Who Have Progressive Disease After First Line Treatment With Checkpoint Inhibitors
Brief Title: Safety and Efficacy of Lenvatinib in Subjects With HCC Progression After First Line Treatment With Checkpoint Inhibitors
Status: Terminated | Type: Observational
Why Stopped: The sponsor withdrawed the sponsorship to the study.
Sponsor: Humanity & Health Medical Group Limited (Other)
Collaborators: Beijing 302 Hospital (Other); Kindai University Faculty of Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: VICI-6
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample for alpha-fetoprotein (AFP) assessment will be obtained by local laboratory every 4 weeks to correlate with each radiographic disease assessment visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lenvatinib: Subjects with HCC progression after first line treatment with checkpoint inhibitors will get the treatment by lenvatinib.
  Interventions: Drug: Lenvatinib
- Non-Lenvatinib: Subjects with HCC progression after first line treatment with checkpoint inhibitors will get the treatment by non-lenvatinib.

INTERVENTIONS:
Drug: Lenvatinib — Prescribed by physician.
  Other Names: Lenvima; E7080
  Groups: Lenvatinib

SUMMARY:
The objective of this study is to evaluate the efficacy of lenvatinib in HCC subjects who have progressive disease after first line treatment with checkpoint inhibitors.

Approximately 20 subjects will be enrollment to evaluate the efficacy and safety of lenvatinib.

CT/MRI assessments will be made at end of first line treatment with checkpoint inhibitors, and every 8-12 weeks thereafter. Disease status will be determined at the site (ie. Investigator and/or radiologist) using RECIST version 1.1.

The primary efficacy endpoint is response rate (RR) defined as proportion of subjects with SD/PR/CR per RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old on the day of consent
2. Capable of understanding and complying with the protocol requirements and signed informed consent
3. Documented histological or cytological diagnosis of HCC
4. HCC progression after first line treatment with checkpoint inhibitors per RECIST 1.1

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Prior TKI treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with HCC progression after first line treatment with checkpoint inhibitors
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | 12 month
  It is the sum of the proportion of stable disease (SD), complete response (CR) and partial response(PR) per RECIST 1.1. That is, RR = SD + CR + PR

SECONDARY OUTCOMES:
Adverse Events | 12 month
  An adverse event (AE) refers to any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, but which does not necessarily have a causal relationship with this treatment. Number and classification of participants with treatment-related adverse events as assessed by CTCAE v4.0 were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanity & Health Clinical Trial Centre, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: No